CLINICAL TRIAL: NCT01567527
Title: 52-week, Multicenter, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy, Safety, and Tolerability of an Intramuscular Depot Formulation of Aripiprazole (OPC-14597) as Maintenance Treatment in Patients With Bipolar I Disorder
Brief Title: Efficacy, Safety, and Tolerability of an Intramuscular Formulation of Aripiprazole (OPC-14597) as Maintenance Treatment in Bipolar I Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Collaborators: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 31-08-250
Record Dates: First submitted 2012-03-26; First posted 2012-03-30 (Estimated); Results first posted 2018-08-24 (Actual); Last update posted 2018-08-24 (Actual); Status verified 2018-07

CONDITIONS: Bipolar I Disorder
Keywords: Aripiprazole; Intramuscular (IM) Depot; Bipolar
MeSH Terms: interventions — Injections, Intramuscular

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Active Comparator: Treatment of Aripiprazole IM Depot
  Interventions: Drug: Intramuscular (IM) Depot Aripiprazole
- 2 (Placebo Comparator): Placebo Comparator: Treatment of IM Depot Placebo
  Interventions: Drug: Intramuscular (IM) Depot Placebo

INTERVENTIONS:
Drug: Intramuscular (IM) Depot Aripiprazole — Formulation: Intramuscular (IM) Depot Aripiprazole Formulation 400 mg or 300 mg, once a month injection
  Arms: 1
Drug: Intramuscular (IM) Depot Placebo — Formulation: Intramuscular (IM) Depot Placebo 400 mg or 300 mg, once a month injection
  Arms: 2

SUMMARY:
This will be a randomized, double-blind, placebo-controlled trial to assess the time to recurrence of any mood episode in subjects with bipolar I disorder who have maintained stability on aripiprazole IM depot for at least 8 weeks. This trial will include male and female subjects 18 to 65 years of age, inclusive, with a diagnosis of bipolar I disorder, according to DSM-IV-TR criteria and confirmed by the Mini International Neuropsychiatric Interview (MINI), who have experienced at least one previous manic episode of sufficient severity to require hospitalization and/or treatment with a mood stabilizer or antipsychotic agent in addition to their current manic episode. All subjects must be experiencing a manic episode (per DSM-IV-TR criteria) with a YMRS total score ≥ 20 at trial entry. Both inpatients and outpatients are eligible for this trial.

This trial will consist of a screening phase followed by 4 treatment phases. Subjects will undergo screening for eligibility, followed by a conversion to oral aripiprazole monotherapy phase, if needed, an oral aripiprazole stabilization phase, a single-blind aripiprazole IM depot stabilization phase, and, a double-blind, placebo-controlled phase.

ELIGIBILITY:
Key Inclusion Criteria:

1. Male and female subjects 18 to 65 years of age, inclusive, at time of informed consent.
2. Subjects with a current diagnosis of bipolar I disorder, as defined by DSM-IV-TR criteria and confirmed by the MINI and a history of at least one previous manic or mixed episode with manic symptoms of sufficient severity to require one of the following interventions: hospitalization and/or treatment with a mood stabilizer, and/or treatment with an antipsychotic agent, in addition to their current manic episode. "Require" is defined as an intervention that occurred rather than one that was recommended. Rapid cyclers with 8 or fewer episodes in the previous year will be included.
3. Subjects currently experiencing a manic episode with a YMRS total score of ≥20 at the Screening Visit.
4. Subjects can have an inpatient or outpatient status prior to entry into Phase C (IM depot stabilization).
5. In the investigator's opinion, subjects who are able to understand the nature of the trial and follow protocol requirements, including the prescribed dosage regimens, tablet ingestion, aripiprazole IM depot injection, and discontinuation of prohibited concomitant medications; who can read and understand the written word in order to complete subject-reported outcomes measures; and who can be reliably rated on assessment scales.

Key Exclusion Criteria:

1. Subjects with a current Axis I (DSM-IV-TR) diagnosis other than bipolar I disorder.
2. Subjects who have NOT experienced at least one previous manic or mixed episode with manic symptoms of sufficient severity to require one of the following interventions: hospitalization and/or treatment with a mood stabilizer, and /or treatment with an antipsychotic agent, excluding their current manic episode. "Require" is defined as a intervention that occurred rather than one that was recommended.
3. Subjects with bipolar I disorder who are considered resistant/refractory to treatment for manic symptoms by history.
4. Subjects unresponsive to clozapine for treatment of mania.
5. Subjects with a significant risk of committing suicide based on history, mental status examination, investigator's judgment, or C-SSRS answer of "yes" to question 4 or 5 (current or within the last 90 days).
6. Subjects with a current manic episode with a duration of > 2 years.
7. Subjects who currently (within the past month) meet DSM-IV-TR criteria for substance abuse or substance dependence; this includes the abuse of alcohol and benzodiazepines, but excludes the use of caffeine and/or nicotine.
8. Subjects who have a history or evidence of a medical condition that would expose them to an undue risk of a significant adverse event (AE) or interfere with assessments of safety or efficacy during the course of the trial, including but not limited to hepatic, renal, respiratory, cardiovascular, endocrine, neurologic, hematologic, or immunologic disease as determined by the clinical judgment of the investigator.
9. Subjects who are currently experiencing a mixed or a depressive episode (per DSM-IV-TR criteria).
10. Subjects with a history of hypersensitivity to antipsychotic agents.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 731 (Actual)
Dates: Start 2012-08; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stacy Wu, MD, Study Director — Otsuka Pharmaceutical Development and Commercialization, Inc.
Locations (76):
- United States (42):
  - Birmingham, Alabama
  - Springdale, Arkansas
  - Beverly Hills, California
  - Costa Mesa, California
  - Escondido, California
  - Garden Grove, California
  - Los Angeles, California
  - National City, California
  - Oceanside, California
  - Orange, California
  - Pico Rivera, California
  - Riverside, California
  - San Diego, California
  - Temecula, California
  - Torrance, California
  - Lauderhill, Florida
  - Leesburg, Florida
  - Melbourne, Florida
  - Oakland Park, Florida
  - Atlanta, Georgia
  - Decatur, Georgia
  - Smyrna, Georgia
  - Hoffman Estates, Illinois
  - New Orleans, Louisiana
  - Rockville, Maryland
  - Flowood, Mississippi
  - Saint Charles, Missouri
  - St Louis, Missouri
  - Lincoln, Nebraska
  - Cherry Hill, New Jersey
  - Brooklyn, New York
  - Buffalo, New York
  - New York, New York
  - Cincinnati, Ohio
  - Dayton, Ohio
  - Oklahoma City, Oklahoma
  - Allentown, Pennsylvania
  - Jenkintown, Pennsylvania
  - Austin, Texas
  - Dallas, Texas
  - Wichita Falls, Texas
  - Richmond, Virginia
- Chatham, Ontario, Canada
- Japan (18):
  - Aizu-Wakamatsu, Fukushima
  - Sapporo, Hokkaido
  - Morioka, Iwate
  - Kawasaki-shi, Kanagawa
  - Yokohama, Kanagawa
  - Kashihara, Nara
  - Sakai, Osaka
  - Sakai-shi, Osaka
  - Fukuoka
  - Itabashi-bu
  - Kanzaki-gun
  - Koriyama-shi
  - Kumamoto
  - Okinawa
  - Shinjuku-ku
  - Tokyo
  - Tottori
  - Toyama
- Poland (4):
  - Gdynia, Pomeranian Voivodeship
  - Bydgoszcz
  - Chełmno
  - Choroszcz
- Romania (3):
  - Târgovişte, Dyambovita
  - Bucharest
  - Judet Lasi
- South Korea (5):
  - Anyang-si, Gyeonggi-do
  - Goyang-si, Gyeonggi-do
  - Daejeon
  - Jeju City
  - Seoul
- Taiwan (3):
  - Keelung
  - Taipei
  - Taouyuan County

REFERENCES:
- [Derived] Calabrese JR, Sanchez R, Jin N, Amatniek J, Cox K, Johnson B, Perry P, Hertel P, Such P, Salzman PM, McQuade RD, Nyilas M, Carson WH. Efficacy and Safety of Aripiprazole Once-Monthly in the Maintenance Treatment of Bipolar I Disorder: A Double-Blind, Placebo-Controlled, 52-Week Randomized Withdrawal Study. J Clin Psychiatry. 2017 Mar;78(3):324-331. doi: 10.4088/JCP.16m11201. PMID 28146613

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial was conducted in 1175 subjects (including 444 screen failures) at 103 trial sites in the following 7 countries: Canada, Japan, Republic of Korea, Poland, Romania, Taiwan, and the United States (US).
Pre-assignment Details: The trial consisted of a screening phase and 4 phases. In Conversion, Oral Stabilization and IM Depot Stabilization Phases, there was a single treatment group. In Double-blind, Placebo-controlled Phase, there were 2 treatment groups. All Outcome Measures were assessed in the Double-blind, Placebo-controlled Phase of the study.
Groups:
- Conversion Phase.: During the Oral Conversion Phase, subjects were cross-titrated from other antipsychotics to oral non-generic aripiprazole monotherapy.
- Oral Aripiprazole Stabilization Phase.: During the Oral Stabilization Phase, subjects were stabilized on an oral dose of aripiprazole. 632 subjects entered the Oral Stabilization Phase (367 subjects entered from the Conversation Phase and 265 subjects entered the Oral Stabilization Phase directly).
- Intramuscular (IM) Depot Stabilization Phase.: During the Depot Stabilization Phase, subjects were stabilized on aripiprazole IM depot. The subjects were assigned to aripiprazole IM depot in the IM Depot Stabilization Phase for a minimum of 12 weeks and a maximum of 28 weeks. To proceed to the Double-blind, Placebo-controlled Phase, subjects were required to meet all the protocol-defined stability criteria for a minimum of 8 consecutive weeks (4 consecutive biweekly visits).
- Double-blind Placebo-controlled Phase - Aripiprazole IM Depot.: Subjects received aripiprazole 300 mg or 400 mg depot intramuscularly up to 52 weeks. A total of 266 subjects entered Double-blind Placebo-controlled phase. Of the 266 subjects, 133 were randomized to aripiprazole IM depot treatment. Since one subject withdrew consent to participate prior to receiving an injection, only 132 subjects received aripiprazole IM depot treatment.
- Double-blind Placebo-controlled Phase - Placebo.: Subjects received placebo intramuscularly up to 52 weeks. A total of 266 subjects entered double-blind placebo-controlled Phase. Of the 266 subjects, 133 were randomized to placebo treatment.
Period: Conversion Phase.
Arm/Group | Conversion Phase. | Oral Aripiprazole Stabilization Phase. | Intramuscular (IM) Depot Stabilization Phase. | Double-blind Placebo-controlled Phase - Aripiprazole IM Depot. | Double-blind Placebo-controlled Phase - Placebo.
Started | 466 | 0 (There were no subjects in this reporting group in this phase of the study.) | 0 (There were no subjects in this reporting group in this phase of the study.) | 0 (There were no subjects in this reporting group in this phase of the study.) | 0 (There were no subjects in this reporting group in this phase of the study.)
Completed | 367 | 0 | 0 | 0 | 0
Not Completed | 99 | 0 | 0 | 0 | 0
Not completed — Protocol deviation | 3 | 0 | 0 | 0 | 0
Not completed — Met withdrawal criteria | 10 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 32 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 16 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 2 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 33 | 0 | 0 | 0 | 0
Not completed — Withdrawn by the investigator | 3 | 0 | 0 | 0 | 0
Period: Oral Aripiprazole Stabilization Phase.
Arm/Group | Conversion Phase. | Oral Aripiprazole Stabilization Phase. | Intramuscular (IM) Depot Stabilization Phase. | Double-blind Placebo-controlled Phase - Aripiprazole IM Depot. | Double-blind Placebo-controlled Phase - Placebo.
Started | 0 (There were no subjects in this reporting group in this phase of the study.) | 632 (265 of the 632 subjects who started this phase entered the Oral Stabilization Phase directly.) | 0 (There were no subjects in this reporting group in this phase of the study.) | 0 (There were no subjects in this reporting group in this phase of the study.) | 0 (There were no subjects in this reporting group in this phase of the study.)
Completed | 0 | 425 | 0 | 0 | 0
Not Completed | 0 | 207 | 0 | 0 | 0
Not completed — Met withdrawal criteria | 0 | 41 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 45 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 44 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 12 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 63 | 0 | 0 | 0
Not completed — Withdrawn by the investigator | 0 | 2 | 0 | 0 | 0
Period: IM Depot Stabilization.
Arm/Group | Conversion Phase. | Oral Aripiprazole Stabilization Phase. | Intramuscular (IM) Depot Stabilization Phase. | Double-blind Placebo-controlled Phase - Aripiprazole IM Depot. | Double-blind Placebo-controlled Phase - Placebo.
Started | 0 (There were no subjects in this reporting group in this phase of the study.) | 0 (There were no subjects in this reporting group in this phase of the study.) | 425 | 0 (There were no subjects in this reporting group in this phase of the study.) | 0 (There were no subjects in this reporting group in this phase of the study.)
Completed | 0 | 0 | 266 | 0 | 0
Not Completed | 0 | 0 | 159 | 0 | 0
Not completed — Protocol deviation | 0 | 0 | 5 | 0 | 0
Not completed — Met withdrawal criteria | 0 | 0 | 26 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 56 | 0 | 0
Not completed — Sponsor discontinued study | 0 | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 21 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 7 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 37 | 0 | 0
Not completed — Withdrawn by the investigator | 0 | 0 | 6 | 0 | 0
Period: Double-blind, Placebo-controlled Phase
Arm/Group | Conversion Phase. | Oral Aripiprazole Stabilization Phase. | Intramuscular (IM) Depot Stabilization Phase. | Double-blind Placebo-controlled Phase - Aripiprazole IM Depot. | Double-blind Placebo-controlled Phase - Placebo.
Started | 0 | 0 | 0 (Subjects were randomized to Aripiprazole IM Depot and placebo groups in this phase of the study) | 133 | 133
Completed | 0 | 0 | 0 | 64 | 38
Not Completed | 0 | 0 | 0 | 69 | 95
Not completed — Protocol deviation | 0 | 0 | 0 | 1 | 1
Not completed — Recurrence of any mood episode with AE | 0 | 0 | 0 | 16 | 33
Not completed — Met withdrawal criteria | 0 | 0 | 0 | 4 | 7
Not completed — AE without recurrence of any moodepisode | 0 | 0 | 0 | 7 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 13 | 10
Not completed — Sponsor discontinued study | 0 | 0 | 0 | 1 | 3
Not completed — Recurrence of any mood episode withoutAE | 0 | 0 | 0 | 19 | 35
Not completed — Lost to Follow-up | 0 | 0 | 0 | 8 | 5

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were presented for the subjects randomized to Double-blind Placebo-controlled Phase. The Double-blind, Placebo-controlled Phase Efficacy Sample consisted of all randomized subjects who received at least 1 injection of IMP and had at least 1 post-baseline efficacy assessment.
Groups:
- Aripiprazole Depot: Subjects received aripiprazole 300 mg or 400 mg depot intramuscularly up to 52 weeks.
- Placebo: Subjects received placebo intramuscularly up to 52 weeks.
- Total: Total of all reporting groups
Arm/Group | Aripiprazole Depot | Placebo | Total
Number analyzed (Participants) | 133 | 133 | 266
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 133 | 132 | 265
  >=65 years | 0 | 1 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.6 (10.8) | 40.6 (11.2) | 40.6 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 83 | 70 | 153
  Male | 50 | 63 | 113
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 2 | 0 | 2
  South Korea | 7 | 7 | 14
  Romania | 8 | 12 | 20
  United States | 101 | 102 | 203
  Japan | 9 | 10 | 19
  Taiwan | 2 | 1 | 3
  Poland | 4 | 1 | 5
Age at first manic episode (years) [Mean (Standard Deviation); unit: years] | 25.2 (10.3) | 24.8 (9.9) | 25.0 (10.1)
Number of mood episodes past 12 months [Mean (Standard Deviation); unit: Mood episodes] | 2.2 (1.2) | 2.2 (1.1) | 2.2 (1.2)
Duration of disease prior to enrollment (years) [Mean (Standard Deviation); unit: years] | 12.1 (9.2) | 13.6 (9.8) | 12.9 (9.5)
Number of prior hospitalizations for a mood episode [Mean (Standard Deviation); unit: Prior hospitalization for mood episode] | 3.5 (3.9) | 3.5 (4.1) | 3.5 (4.0)
Young-Mania Rating Scale (YMRS) Total Score [Mean (Standard Deviation); unit: Scores on a scale] — The YMRS consisted of 11 items to assess the core symptoms of mania. Four items (irritability, speech, content, and disruptive-aggressive behavior) were graded on a scale of 0 to 8 (a higher score indicated increased severity) and 7 items (elevated mood, increased motor activity/energy, sexual interest, sleep, language-thought disorder, appearance, and insight) were graded on a scale of 0 to 4 (a higher score indicated increased severity). The scores from 11 items were summed to a total score ranging from 0 to 60 (higher score indicated greater severity of symptoms).
  Scores on a scale | 2.9 (3.5) | 2.6 (3.0) | 2.8 (3.3)
Montgomery Asberg Depression Rating Scale (MADRS) Total Score [Mean (Standard Deviation); unit: Scores on a scale] — The MADRS measured the depression level of a participant. This scale consisted of 10 items (reported sadness, apparent sadness, inner tension, reduced sleep, reduced appetite, concentration difficulties, lassitude, inability to feel, pessimistic thoughts, and suicidal thoughts), each with 7 defined grades of severity graded on a scale of 0 to 6 (a higher score indicated increased severity) . The overall total score was 0 to 60; 0, no depression; 60, severely depressed. The missing score for any one item resulted in a missing MADRS total score.
  Scores on a scale | 3.0 (3.4) | 2.4 (3.4) | 2.7 (3.4)
Clinical Global Impressions - Bipolar Version Severity (CGI-BP-S) - Mania [Mean (Standard Deviation); unit: Scores on a scale] — CGI-BP-S assessed the subject's severity of Illness (mania) based on a 7-point scale ranging from 1 (normal/ not ill at all) to 7 (very severely ill).
  Scores on a scale | 1.5 (0.7) | 1.4 (0.6) | 1.5 (0.7)

OUTCOME MEASURES:

1. Primary Outcome: Time From Randomization to Recurrence of Any Mood Episode During Double-bind Placebo-controlled Phase.
Description: This endpoint was defined as meeting any of the following criteria:
  1. Hospitalization for any mood episode OR
  2. Any of the following:
     1. YMRS total score ≥ 15 OR
     2. MADRS total score ≥ 15 OR
     3. CGI-BP-S score > 4 (overall score) OR
  3. SAE of worsening disease (bipolar I disorder) OR
  4. Discontinuation due to lack of efficacy or discontinuation due to an AE of worsening disease OR
  5. Clinical worsening with the need for treatment of symptoms of an underlying mood disorder by addition of a mood stabilizer, antidepressant treatment, antipsychotic medication, or increase greater than the allowed benzodiazepine doses, or
  6. Active suicidality, which is defined as a score of 4 or more on the MADRS item 10 OR an answer of "yes" on question 4 or 5 on the C-SSRS.
  The time to event is presented in the following table.
Time Frame: Baseline of the Double-blind, Placebo-controlled Phase Up to the end of the study (Week 52).
Population: All randomized subjects who received at least one injection of investigational medicinal product (IMP) and had at least one post-baseline efficacy assessment in the Double-blind, Placebo-controlled Phase, eg, modified intent-to-treat (ITT) population.
Measure: Median (95% Confidence Interval); unit: Days
Groups:
- Aripiprazole IM Depot: Subjects received aripiprazole 300 mg or 400 mg depot intramuscularly up to 52 weeks.
Arm/Group | Aripiprazole IM Depot | Placebo
Number analyzed (Participants) | 132 | 133
Days | NA [NA to NA] — Here NA means values which were not estimable. The values for median and its 95% confidence interval of time to recurrence were not estimable due to the number of subjects with event was low. | 308 [178 to NA] — Here NA means values which were not estimable. The upper limit of 95% confidence interval of time to recurrence was not estimable in Placebo arm due to the number of subjects with event was low.
Statistical Analysis 1: Comparison: Aripiprazole IM Depot vs Placebo; Significance level 0.05; Test type: Superiority; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.451, 95% CI 2-sided [0.299 to 0.678] — Using the Cox proportional hazards model with term for treatment group. HR is estimated for Aripiprazole IM depot relative to Placebo
Statistical Analysis 2: Comparison: Aripiprazole IM Depot vs Placebo; Test type: Superiority — Using the Cox proportional hazards model with term for treatment group; Hazard Ratio (HR) = 2.22, 95% CI 2-sided [1.475 to 3.34] — HR is estimated for Placebo relative to Aripiprazole IM depot

2. Secondary Outcome: Number of Subjects Meeting Criteria for Recurrence of Any Mood Episode.
Description: To assess the proportion of subjects who met criteria for recurrence of any mood episode (manic, mixed or depressive). Hierarchical procedure was used to preserve the overall Type I error at 0.05.
Time Frame: Baseline of the Double-blind, Placebo-controlled Phase Up to the end of the study (Week 52).
Population: All randomized subjects who received at least one injection of IMP and had at least one post-baseline efficacy assessment in the Double-blind, Placebo-controlled Phase, eg, modified ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | Aripiprazole IM Depot | Placebo
Number analyzed (Participants) | 132 | 133
Participants | 35 | 68
Statistical Analysis 1: Comparison: Aripiprazole IM Depot vs Placebo; Statistical analysis for any mood episode; Test type: Superiority — Using a hierarchical procedure to preserve the overall Type I error rate at 0.05, after testing the primary outcome; p < 0.0001, Fisher Exact; Percentage Difference (Final Values) = -24.6, 95% CI 2-sided [-36.7 to -12.5]

3. Secondary Outcome: Mean Change From Randomization to Endpoint in the CGI-BP-S (Mania) Score.
Description: CGI-BP-S assessed the subject's severity of Illness (mania) based on a 7-point scale ranging from 1 (normal/ not ill at all) to 7 (very severely ill).
Time Frame: Baseline of the Double-blind, Placebo-controlled Phase up to the end of the study (Week 52).
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Aripiprazole IM Depot | Placebo
Number analyzed (Participants) | 131 | 133
Units on a scale | -0.16 (0.058) | 0.27 (0.126)
Statistical Analysis 1: Comparison: Aripiprazole IM Depot vs Placebo; Test type: Superiority — Using mixed model repeated measures (MMRM) analysis with a restricted maximum likelihood (REML) approach. Analyses included the categorically fixed effects of treatment, region, trial week, and treatment-by-week interaction, as well as the continuously fixed covariates of baseline-score-by-week interaction. An unstructured covariance structure was used to model the within-subject errors and Kenward-Rodger degree of freedom was used to test the fixed effects; p = 0.0011, Mixed model repeated measure analysis; Mean Difference (Final Values) = -0.43, 95% CI 2-sided [-0.69 to -0.17]

4. Secondary Outcome: Time From Randomization to Recurrence Defined by Hospitalization for a Mood Episode.
Description: Analysis of time from randomization to recurrence defined by hospitalization for a mood episode (Double-blind, Placebo-controlled Phase efficacy sample).
  Time to recurrence is presented in the following table.
Time Frame: Baseline of the Double-blind, Placebo-controlled Phase up to the end of the study (Week 52).
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Aripiprazole IM Depot | Placebo
Number analyzed (Participants) | 132 | 133
Days | NA [NA to NA] — Here NA means values which were not estimable. The values for median and its 95% confidence interval of time to recurrence were not estimable due to the number of subjects with event was low. | NA [NA to NA] — Here NA means values which were not estimable. The values for median and its 95% confidence interval of time to recurrence were not estimable in Placebo arm due to the number of subjects with event was low.
Statistical Analysis 1: Comparison: Aripiprazole IM Depot vs Placebo; Test type: Superiority; p = 0.0002, Log Rank; Hazard Ratio (HR) = 0.137, 95% CI 2-sided [0.04 to 0.465] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Aripiprazole IM Depot vs Placebo; Test type: Superiority — Using the Cox proportional hazards model with term for treatment group; Hazard Ratio (HR) = 7.313, 95% CI 2-sided [2.151 to 24.865] — HR is estimated for Placebo relative to Aripiprazole IM depot

ADVERSE EVENTS:
Time Frame: Any AEs were recorded from the signing of informed consent up to 52 weeks (end of the study).
Description: Safety analysis set (SAF): The SAF included all subjects who received at least one dose of trial medication in all phases of the study. Safety analysis results were reported for the safety populations.
Groups:
- Conversion Phase.: During the Oral Conversion Phase, subjects were cross-titrated from other antipsychotics to oral non-generic aripiprazole monotherapy. Received Oral aripiprazole at a target starting dose of 15 mg/day.
- Oral Aripiprazole Stabilization Phase.: Subjects received oral aripiprazole dose ranging from 15 mg to 30 mg daily.
- IM Depot Stabilization Phase.: During the depot stabilization phase, subjects were stabilized on aripiprazole depot.
- Aripiprazole IM Depot- Double-blind, Placebo-controlled Phase.: Subjects received IM depot aripiprazole 400 mg or 300 mg, once a month injection.
- Placebo-Double-blind, Placebo-controlled Phase.: Subjects received IM Depot Placebo, once a month injection.
Arm/Group | Conversion Phase. | Oral Aripiprazole Stabilization Phase. | IM Depot Stabilization Phase. | Aripiprazole IM Depot- Double-blind, Placebo-controlled Phase. | Placebo-Double-blind, Placebo-controlled Phase.
All-Cause Mortality (participants affected / at risk) | 0/459 | 1/614 | 0/425 | 1/132 | 0/133
Serious Adverse Events (participants affected / at risk) | 32/459 | 35/614 | 36/425 | 10/132 | 25/133
Other Adverse Events (participants affected / at risk) | 180/459 | 196/614 | 194/425 | 66/132 | 62/133
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Conversion Phase. (N=459) | Oral Aripiprazole Stabilization Phase. (N=614) | IM Depot Stabilization Phase. (N=425) | Aripiprazole IM Depot- Double-blind, Placebo-controlled Phase. (N=132) | Placebo-Double-blind, Placebo-controlled Phase. (N=133)
Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Akathisia (Nervous system disorders) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Brain injury (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Radiculopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Affect lability (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Affective disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aggression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bipolar disorder (Psychiatric disorders) | 6 (6) | 2 (2) | 0 (0) | 1 (1) | 3 (3)
Bipolar I disorder (Psychiatric disorders) | 4 (4) | 1 (1) | 4 (4) | 2 (2) | 3 (3)
Hypomania (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Major depression (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Mania (Psychiatric disorders) | 13 (14) | 17 (17) | 7 (7) | 2 (2) | 10 (10)
Suicide attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depressed mood (Psychiatric disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 4 (4) | 8 (8) | 0 (0) | 0 (0)
Depressive symptom (Psychiatric disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 2 (2) | 3 (3) | 3 (3) | 0 (0) | 0 (0)
Colitis ulcerative (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pelvic adhesions (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vulval abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute Kidney Injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal Tubular Necrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Extrapyramidal disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Conversion Phase. (N=459) | Oral Aripiprazole Stabilization Phase. (N=614) | IM Depot Stabilization Phase. (N=425) | Aripiprazole IM Depot- Double-blind, Placebo-controlled Phase. (N=132) | Placebo-Double-blind, Placebo-controlled Phase. (N=133)
Weight increased (Investigations) | 13 (13) | 22 (23) | 47 (47) | 31 (31) | 24 (25)
Akathisia (Nervous system disorders) | 76 (84) | 94 (99) | 74 (82) | 27 (32) | 17 (20)
Headache (Nervous system disorders) | 31 (64) | 13 (21) | 12 (12) | 4 (4) | 9 (10)
Fatigue (General disorders) | 14 (14) | 19 (19) | 22 (25) | 4 (4) | 5 (6)
Anxiety (Psychiatric disorders) | 19 (20) | 24 (24) | 30 (36) | 9 (9) | 6 (6)
Insomnia (Psychiatric disorders) | 35 (37) | 34 (35) | 41 (47) | 10 (11) | 10 (12)
Restlessness (Psychiatric disorders) | 36 (45) | 32 (34) | 24 (25) | 6 (6) | 5 (5)
Nasopharyngitis (Infections and infestations) | 18 (18) | 11 (11) | 22 (30) | 10 (13) | 13 (29)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Until the information herein is released by Otsuka to the public domain, the contents of this document are Otsuka confidential information and should not be duplicated or re-distributed without prior written consent of Otsuka.